CLINICAL TRIAL: NCT06287424
Title: An Exploratory Eighteen Month Clinical Study To Evaluate Efficacy Of AGE Product On Periodontitis, A Dose Response Study
Brief Title: The Efficacy Of AGE On Periodontitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hadassah Medical Organization (Other)
Collaborators: Wakunaga Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: HMO-2O-0536
Record Dates: First submitted 2021-03-09; First posted 2024-03-01 (Actual); Last update posted 2024-03-01 (Actual); Status verified 2021-03

CONDITIONS: Periodontitis
Keywords: Garlic; Periodontitis; Gingival Bleeding
MeSH Terms: conditions — Periodontitis; Gingival Hemorrhage

STUDY DESIGN:
Intervention Model Description: 4 Regimen parralel groups
Who Masked: Participant
Masking Description: Eligible subjects will be stratified based on Screening mean PPD (above or below 2mm), mean GBI (above or below 0.44), mean age (above or below 45 years old), gender (male or female) and tobacco use (yes or no). Within strata, subjects will be randomly assigned to one of the treatment groups using an encoded program. This assignment process and the distribution of test products will be conducted in a protected area that will ensure blinding of the examiner to the identity of the test products.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- A: 4 tablet per day (Experimental): • Group A: Daily use of Aged Garlic Extract product: Take two (2) tablets with a meal twice daily.
  The label is:
  Garlic extract tablets for research - for research use only Instructions for use: Take (2) tablets immediately after breakfast and (2) tablets immediately after dinner every day.
  Storage: Store in a cool, dry place with the lid tightly closed. Expiration date: August 2022 Please return empty bottles and excess tablets as requested.
  Interventions: Dietary Supplement: Aged Garlic Extract
- B: 6 tablet per day (Experimental): • Group B: Daily use of Aged Garlic Extract product: Take three (3) tablets with a meal twice daily.
  The label is:
  Garlic extract tablets for research - for research use only Instructions for use: Take (3) tablets immediately after breakfast and (3) tablets immediately after dinner every day.
  Storage: Store in a cool, dry place with the lid tightly closed. Expiration date: August 2022 Please return empty bottles and excess tablets as requested.
  Interventions: Dietary Supplement: Aged Garlic Extract
- C: 8 tablet per day (Experimental): • Group C: Daily use of Aged Garlic Extract product: Take four (4) tablets with a meal twice daily.
  The label is:
  Garlic extract tablets for research - for research use only Instructions for use: Take (4) tablets immediately after breakfast and (4) tablets immediately after dinner every day.
  Storage: Store in a cool, dry place with the lid tightly closed. Expiration date: August 2022 Please return empty bottles and excess tablets as requested.
  Interventions: Dietary Supplement: Aged Garlic Extract
- D: Placebo (Placebo Comparator): • Group C: Daily use of Aged Garlic Extract product: Take four (4) tablets with a meal twice daily.
  The label is:
  Garlic extract tablets for research - for research use only Instructions for use: Take (4) tablets immediately after breakfast and (4) tablets immediately after dinner every day.
  Storage: Store in a cool, dry place with the lid tightly closed. Expiration date: August 2022 Please return empty bottles and excess tablets as requested.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Aged Garlic Extract — Subjects will be instructed to continue using their regular home oral hygiene products until the Product Distribution Visit (Visit 2). They will also be instructed not to add or change any of their regular home oral hygiene products during that time.
  Arms: A: 4 tablet per day; B: 6 tablet per day; C: 8 tablet per day
Dietary Supplement: Placebo — Placebo
  Arms: D: Placebo

SUMMARY:
The objective of this study is to assess the long-term efficacy of "AGE among on deep periodontal pockets by different doses of "AGE" for a period of 18 months.

DETAILED DESCRIPTION:
This is a randomized, controlled, examiner-blind, 4-treatment parallel group study. The study will be conducted at the Hebrew University, Hadassah, Israel. A sufficient number of subjects will be screened to obtain approximately 300 generally healthy adult volunteers with moderate to deep periodontal pockets.

Subjects will be stratified and randomly assigned equally to either one from the 3 regimen groups with different doses of AGE or a control group (Placebo).

Subjects will be requested to use the products at home for the duration of the study according to the written and verbal usage instructions given to them during product distribution. At Baseline, Month 6, Month 12, and Month 18, subjects will receive oral soft tissue exams, and will have periodontal measurements made as described in below.

All groups will receive supra-gingival dental prophylaxes every 6 month consistent with local norms and standards. Products will be re-supplied approximately every six months following Baseline. During study conduct, subjects with evidence of progressive periodontal disease (≥3 mm increases in pocket depth, attachment loss or recession) will be exited from the study and treated following local norms.

ELIGIBILITY:
Inclusion Criteria:

* give written informed consent and receive a copy of their consent;
* be between the ages of 30-60 years;
* be in good general health as determined by the Investigator/designee based on a review of the medical history/update for participation in the study;
* possess a minimum of 16 natural teeth (excluding third molars) with facial and lingual scorable surfaces;
* have at least 20 bleeding sites (sum of sites with a score of 1 or 2 on the GBI index);
* have at least: 3 eligible periodontal pockets sites (PPD 3.5-6 mm, bleeding);
* agree to delay any elective dentistry until study completion, including additional dental prophylaxes outside the study protocol;
* agree to refrain from using any non-study oral hygiene products for the study duration (subject will be allowed to continue using floss but they will be instructed not to add/change any other oral hygiene products, including whitening products etc);
* agree not to participate in any other oral care clinical study for the duration of this study;
* agree to return for their scheduled visits and follow study procedures;

Exclusion Criteria:

* • severe periodontal disease, as characterized by purulent exudate, generalized mobility, and/or a new severe recession;

  * active treatment for periodontitis;
  * having a medical condition requiring antibiotic pre-medication prior to dental procedures,
  * fixed facial or lingual orthodontic appliances or removable partial dentures;
  * antibiotic or chlorhexidine use or anti-inflammatory medications within two weeks prior to Screening visit;
  * self-report nursing, pregnancy, or intent to become pregnant during the study;
  * dental prophylaxis within two month prior to the Screening visit;
  * any diseases or conditions that could be expected to interfere with the subject safely completing the study;

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 300 (Actual)
Dates: Start 2021-04-04 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2023-01-01 (Actual)

PRIMARY OUTCOMES:
Gingival Bleeding Index (GBI) | Baseline, 6 Month, 12 Month, 18 Month
  The gingiva should be lightly air-dried and a periodontal probe with a 0.5 mm diameter tip inserted into the gingival crevice to a depth of 2mm or until slight resistance is felt. The probe is then run gently around the tooth at an angle of approximately 60° and in contact with the sulcular epithelium. Minimum axial force is used to avoid undue penetration into the tissue and the probe is moved around the crevice, gently stretching the epithelium. Each of the 3 gingival areas, i.e., buccal, mesial and lingual, of the teeth will be probed in this manner waiting approximately 30 seconds before recording the number of gingival units which bleed
Probing Pocket Depth (PPD) | Baseline, 12 Month, 18 Month
  Probing Pocket Depth at every site will be assessed as the distance from the gingival margin to the apical end of the pocket using a WHO CPI probe. The probe will be inserted parallel to the root surface and directed apically toward the perceived location of the apex of the root until slight resistance is felt. Probe recordings will be rounded off to the nearest millimeter mark.

CONTACTS AND LOCATIONS:
Locations (1):
- Hebrew University, Jerusalem, Israel

IPD SHARING:
Plan to Share IPD: No